CLINICAL TRIAL: NCT00218010
Title: Breastfeeding Among Methadone Maintained Women
Brief Title: Methadone Levels in Breast Milk of Women Taking Methadone for Opiate Addiction - 2
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Associate Professor of Pediatrics, National Institute on Drug Abuse (NIDA)
Other Study IDs: NIDA-00495-2
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2015-04

CONDITIONS: Breast Feeding; Opioid-Related Disorders
Keywords: methadone; lactation; breastfeeding; maternal opioid dependency
MeSH Terms: conditions — Breast Feeding; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Methadone maintained lactating women: Methadone maintained women who chose to breastfeed their infants provided breast milk and plasma samples for this study.

SUMMARY:
Methadone is a drug that offers significant therapeutic benefits to opiate dependent women who are pregnant. Currently, it is the treatment of choice for this group of people. The purpose of this study is to determine the amount of methadone in the breast milk of women who are breastfeeding and taking methadone for opiate addiction. In addition, this study will evaluate the effects of methadone on infant neurobehavior.

DETAILED DESCRIPTION:
Methadone is a drug that is commonly used to treat opiate addiction, usually as part of a detoxification and maintenance program. Methadone offers significant therapeutic benefits to pregnant women who are opiate dependent, and it is currently the treatment of choice for this group of people. In general, breast milk is beneficial for infants. However, there is some concern as to whether it is safe for women who are taking methadone to breastfeed their babies. The purpose of this study is to determine the amount of methadone in the breast milk of women who are breastfeeding and taking methadone for opiate addiction. In addition, this study will evaluate the effects of methadone on infant neurobehavior.

Participants will be assigned to one of two groups: women taking methadone who will breastfeed their babies or women taking methadone who will bottle-feed their babies. On Days 1, 2, 3, 4, 14, and 30, following infant delivery, plasma will be collected from both groups and breast milk will be collected from the breastfeeding group. These samples will be quantitatively analyzed for methadone. Infants will undergo neurobehavioral assessments on Days 3, 14, and 30, following birth. Rates and severity of neonatal abstinence syndrome will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy methadone-maintained women electing to either exclusively breastfeed or bottle-feed their infants for 1 month after delivery

Exclusion Criteria:

* Relapse to illicit drugs or alcohol at any time during the study
* Positive maternal or infant urine toxicology test at birth
* Serious medical or psychiatric illness requiring medication or medical intervention
* HIV infected
* Currently dependent on alcohol
* Major birth defect in the infant
* Significant medical problems in the infant, including premature birth, sepsis, or other infections

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: lactating women
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2000-11; Primary Completion 2005-08 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
methadone concentrations in breast milk | 1-30 days after delivery
methadone concentrations in maternal plasma | 1-30 days after delivery

SECONDARY OUTCOMES:
methadone concentrations in infant plasma | 1-30 days after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M. Jansson, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University (BPRU) Bayview Campus, Baltimore, Maryland, United States

REFERENCES:
- [Background] Jansson LM, Velez M, Harrow C. Methadone maintenance and lactation: a review of the literature and current management guidelines. J Hum Lact. 2004 Feb;20(1):62-71. doi: 10.1177/0890334403261027. PMID 14974702
- [Result] Jansson LM, Choo R, Velez ML, Lowe R, Huestis MA. Methadone maintenance and long-term lactation. Breastfeed Med. 2008 Mar;3(1):34-7. doi: 10.1089/bfm.2007.0032. PMID 18333767
- [Result] Jansson LM, Choo R, Velez ML, Harrow C, Schroeder JR, Shakleya DM, Huestis MA. Methadone maintenance and breastfeeding in the neonatal period. Pediatrics. 2008 Jan;121(1):106-14. doi: 10.1542/peds.2007-1182. PMID 18166563
- [Result] Jansson LM, Choo RE, Harrow C, Velez M, Schroeder JR, Lowe R, Huestis MA. Concentrations of methadone in breast milk and plasma in the immediate perinatal period. J Hum Lact. 2007 May;23(2):184-90. doi: 10.1177/0890334407300336. PMID 17478871